CLINICAL TRIAL: NCT07003412
Title: The PULSE PVC Registry Evaluates the Safety and Efficacy of Focal PFA Using the Centauri System for Symptomatic PVCs Across European Centers, With Outcomes Stratified by Site of Origin and Compared to Historical RF Ablation Data.
Brief Title: PULSE PVC Registry: Multicenter Study on Focal Pulsed Field Ablation for Premature Ventricular Contractions
Status: Enrolling by invitation | Type: Observational
Sponsor: Zentralklinik Bad Berka (Other)
Responsible Party: Principal Investigator, Ahmad Keelani, Principal Investigator, Zentralklinik Bad Berka
Other Study IDs: 23333/2024/62
Record Dates: First submitted 2025-05-18; First posted 2025-06-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Premature Ventricular Contraction (PVC); Pulsed Field Ablation
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PULSE PVC Registry is a European multicenter observational study designed to assess the safety and efficacy of focal pulsed field ablation (PFA) using the Centauri Generator system in patients with symptomatic premature ventricular contractions (PVCs). The registry collects standardized procedural and follow-up data across diverse PVC origins, enabling comparisons with historical radiofrequency (RF) ablation outcomes. Data will include baseline characteristics, procedural details, complications, and long-term PVC burden reduction. Each center will obtain local ethics approval, and only anonymized data will be analyzed.

DETAILED DESCRIPTION:
The PULSE PVC Registry is a European multicenter observational registry designed to evaluate the safety, feasibility, and midterm outcomes of focal pulsed field ablation (PFA) for the treatment of symptomatic premature ventricular contractions (PVCs). The study includes patients undergoing focal PFA using a monopolar biphasic energy system (Centauri Generator), across multiple high-volume electrophysiology centers in Europe.

The registry collects detailed baseline demographics, comorbidities (e.g., hypertension, diabetes, chronic kidney disease), structural heart disease status, antiarrhythmic drug use, prior ablation history, and baseline PVC burden. Procedural characteristics include PVC mapping approach, pharmacologic testing (e.g., isoproterenol, nitroglycerin), number and type of ablation applications (PFA and/or RF), use of coronary angiography, venous system access (GCV/AIV), and fluoroscopy metrics.

Outcomes assessed include:

Primary outcome: Midterm clinical success, defined as a reduction in PVC burden to <5% on follow-up (via Holter monitoring)

Secondary outcomes: Acute procedural success, complication rates (e.g., coronary vasospasm, conduction disturbances, stroke, vascular complications), and recurrence patterns.

Patients are stratified based on the site of origin of PVCs (e.g., RVOT subregions, LVOT, aortic cusps, papillary muscles).

Follow-up includes symptom assessment, PVC burden, antiarrhythmic drug use, and mode of follow-up (telephone or in-person). The registry provides a comprehensive overview of clinical outcomes with focal PFA and enables comparison with historical radiofrequency ablation data.

This registry aims to generate robust real-world evidence to inform procedural strategy, patient selection, and safety considerations in PVC ablation using pulsed field energy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic PVCs who underwent focal monopolar biphasic PFA
* Use of Centauri Generator system
* Minimum 3-month clinical follow-up at time of data entry

Exclusion Criteria:

* Incomplete procedural or follow-up data
* Patients receiving exclusively RF ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: he study population consists of adult patients (age ≥18 years) with symptomatic premature ventricular contractions undergoing focal monopolar biphasic pulsed field ablation. All patients included must have been treated with the Centauri Generator system and have a minimum of 3 months of follow-up data available at the time of registry entry. The population is expected to be heterogeneous, including patients with and without structural heart disease, and PVCs originating from various anatomical sites. Patients will be enrolled across multiple European electrophysiology centers with varying procedural practices, enhancing the generalizability of the findings.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically significant PVCs at 6-month follow-up | through study completion, an average of 6 months
  Clinically significant PVCs are defined as a PVC burden ≥5% on 24-hour Holter ECG. The primary efficacy endpoint is the proportion of patients who achieve a reduction in PVC burden to <5% at 6 months following pulsed field ablation (PFA). PVC burden will be quantified using standardized 24-hour Holter recordings. Patients must not be on any new antiarrhythmic medication during this period to be considered a true efficacy responder.

SECONDARY OUTCOMES:
Acute Procedural Success | Day 0 to Day 2 (during hospital stay)
  Acute procedural success is defined as complete elimination of the targeted PVC morphology by the end of the ablation procedure, confirmed by the absence of spontaneous or inducible PVCs following programmed stimulation and/or isoproterenol challenge.
  Early PVC burden reduction is assessed via telemetry and 24-hour Holter monitoring performed during hospitalization. A PVC burden <5% during the first 48 hours post-ablation is considered an early indicator of treatment efficacy.
Periprocedural Complication Rate | Day 0 to Day 2 (hospital stay)
  Procedure-related complications occurring during the hospital stay will be systematically recorded from the end of the procedure until discharge (typically Day 0 to Day 2). These include vascular complications (e.g., access-site hematoma, iliac artery dissection), conduction disturbances (e.g., transient or persistent right bundle branch block), coronary vasospasm, and cerebrovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: J. Christoph Geller, Prof. Dr., Study Director — Zentralklinikum Bad berka; Santi Raffa, Dr., Study Director — Zentralklinik Bad Berka
Locations (1):
- Zentralklinik Bad Berka, Bad Berka, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding IPD sharing is currently under review and will depend on institutional policies, ethical approvals.